CLINICAL TRIAL: NCT05617417
Title: Evaluation of the Efficacy of Locally Administered Autologous Injectable Platelet-rich Fibrin in Women With Stress Urinary Incontinence
Brief Title: The Efficacy of Injectable Platelet-rich Fibrin in the Treatment of the Female Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ulku Mete Ural, Professor Doctor, Abant Izzet Baysal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAIBU-MF-OG-UMU-001
Record Dates: First submitted 2022-10-25; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Urinary Incontinence; Treatment
Keywords: Urinary Stress Incontinence; Platelet-Rich Fibrin; Questionnaire
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Thirty patients with pure stress urinary incontinence were included in the study. Autologously prepared injectable platelet-rich fibrin from the patients was applied locally. The procedure was repeated for the same patient three times with an interval of one month. The severity of urinary incontinence was evaluated and recorded by filling out questionnaires before and after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The women with stress urinary incontinence administered injectable platelet-rich fibrin (Other): Injectable platelet-rich fibrin was prepared by centrifuging venous blood samples from women with stress urinary incontinence. The obtained autologous material was injected into the anterior vaginal wall, approximately 1.5 cm below the urethral meatus, without applying a local anesthetic. The procedure was repeated for the same patient three times with an interval of one month. The severity of urinary incontinence was evaluated by filling out questionnaires before and after the procedure.
  Interventions: Other: Local applied injectable platelet-rich fibrin in women with stress urinary incontinence

INTERVENTIONS:
Other: Local applied injectable platelet-rich fibrin in women with stress urinary incontinence — Injectable platelet-rich fibrin was prepared by centrifuging venous blood taken from women with stress urinary incontinence and applied locally to the anterior vaginal wall of the patients.

SUMMARY:
We aimed to evaluate the efficacy of locally applied injectable platelet-rich fibrin in women with stress urinary incontinence. We searched whether there was a decrease in the severity of urinary incontinence after the injection of platelet-rich fibrin.

The participants will answer questionnaires about urinary incontinence before and after the injectable platelet-rich fibrin treatment.

DETAILED DESCRIPTION:
Female patients with pure stress urinary incontinence who gave written informed consent after being informed about the study were included in the study. Two tubes of venous blood samples taken from the patients were centrifuged and injectable platelet-rich fibrin was prepared. The obtained autologous material was injected into the patient within one minute after preparation, without applying a local anesthetic. The injection was given to the anterior wall of the vagina, approximately 1.5 cm below the urethral meatus, coinciding with the mid-urethral region, and the dose was applied to three adjacent points. The procedure was repeated three times at one-month intervals. Before and after the procedure, ICIQ-SF, UDI-6, and IIQ-7 questionnaires were filled and the severity of urinary incontinence was recorded.

ELIGIBILITY:
Inclusion Criteria:

* The patient who has pure stress urinary incontinence

Exclusion Criteria:

* The patient who had previous surgery for stress urinary incontinence
* Known platelet dysfunction
* Anti-coagulant users
* Critical thrombocytopenia

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Changes in urinary incontinence severity before and 6 months after injectable platelet-rich fibrin application were evaluated with International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF). | Change in urinary incontinence severity before and 6 months after treatment
  ICIQ-SF evaluates the severity of urinary incontinence symptoms and their impact on health-related quality of life. It is scored on a scale from 0-21. A higher score indicates greater impairment from incontinence. Stress urinary incontinence grade according to ICIQ-SF: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21).

SECONDARY OUTCOMES:
Changes in quality of life in patients with urinary incontinence before and 6 months after injectable platelet-rich fibrin application were evaluated with Urogenital Distress Inventory-6 (UDI-6) and Incontinence Impact Questionnaire-7 (IIQ-7). | Change in urinary incontinence severity before and 6 months after treatment
  UDI-6 is a short version of a condition-specifc quality of life instrument. Higher scores in UDI-6 indicate higher disability. Total score is from 0 to 100.
  IIQ-7 is a urinary incontinence-specific psychometric questionnaire. This questionnaire assesses the psychosocial impact of UI in women. Higher scores in UDI-6 indicate higher disability. Total score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü Mete Ural, Principal Investigator — Bolu Abant Izzet Baysal University, Faculty of Medicine, Department of Obstetrics and Gynecology
Locations (1):
- Bolu Abant Izzet Baysal University, Faculty of Medicine, Bolu, Gölköy, Turkey (Türkiye)